CLINICAL TRIAL: NCT00780663
Title: A Phase 2, Multi-Center, Open Label Study Evaluating the Efficacy and Safety of Quarfloxin in Patients With Low to Intermediate Grade Neuroendocrine Carcinoma
Brief Title: Quarfloxin in Patients With Low to Intermediate Grade Neuroendocrine Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cylene Pharmaceuticals (Industry)
Responsible Party: Claire Padgett, VP Clinical Operations, Cylene Pharmaceuticals Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C3-07-003
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Neuroendocrine Tumors; Carcinoid Tumor
Keywords: Neuroendocrine; Carcinoid; NET; MEN-1; Islet cell
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoid Tumor | interventions — CX 3543

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Quarfloxin (Experimental): Single arm study - open label.
  Interventions: Drug: Quarfloxin

INTERVENTIONS:
Drug: Quarfloxin — IV Quarfloxin 240 mg/m2 daily x5 days every 21 days
  Other Names: CX-3543

SUMMARY:
This is a Phase 2, open-label, multicenter, efficacy and safety study of quarfloxin in patients with low or intermediate grade neuroendocrine cancer. The purpose of this study is to evaluate the rate of clinical benefit response to quarfloxin treatment including the reduction in secretory symptoms of flushing and/or diarrhea or the reduction quantifiable hormones or other biochemical tumor markers.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed low or intermediate grade neuroendocrine carcinoma including carcinoid and islet cell cancer. Patients with neuroendocrine tumors associated with MEN1 syndrome are eligible.
* Measureable disease by RECIST
* Unresectable or metastatic disease
* Secretory symptoms of diarrhea or flushing or both attributed to their carcinoid tumor and/or quantifiable hormones or other biochemical markers
* Males and females 18 years of age or older.
* Zero to two prior cytotoxic chemotherapy regimens.
* Patients may be receiving concomitant octreotide Sandostatin®
* Patients must have central IV access, or agree to the insertion of a central IV line.
* All previous cancer therapies, radiation, and surgery, must have been discontinued at least 21 days prior to the start of treatment.
* Acceptable liver function
* Acceptable renal function
* Acceptable hematologic status
* ECOG Performance Status ≤1.
* Anticipated survival of at least 6 months.
* Able to maintain a patient diary.
* For men and women of child-producing potential, use of effective contraceptive methods during the study and for one month after discontinuation of treatment.
* Ability to understand the requirements of the study, provide written informed consent and agree to abide by the study restrictions and return to the clinic for required assessments.

Exclusion Criteria:

* Poorly differentiated neuroendocrine carcinoma, high-grade neuroendocrine carcinoma, adenocarcinoid, goblet cell carcinoid or small cell carcinoma.
* Pregnant or nursing women.
* Severe chronic obstructive pulmonary disease with hypoxemia or an uncorrectable pulmonary compromise.
* Seizures not controlled by anticonvulsant therapy.
* Participation in any investigational drug study within 28 days before quarfloxin administration or currently receiving investigational therapy.
* Patients with a second malignancy requiring active treatment.
* Active symptomatic bacterial, fungal, or viral infection including active HIV or viral hepatitis.
* Prior treatment with quarfloxin.
* Clinically significant bleeding event within the last 3 months, unrelated to trauma, or underlying condition that would be expected to result in a bleeding diathesis.
* Patients who have exhibited allergic reactions to a similar structural compound or formulation.
* Any illness or condition that in the opinion of the investigator may affect safety of treatment or evaluation of any of the study's endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Clinical benefit. Clinical benefit is defined as a reduction of secretory symptoms or reduction of quantifiable hormones or other biochemical tumor markers where concomitantly there is an absence of radiological evidence for tumor progression. | monthly for clinical benefit, every two months for tumor progression

SECONDARY OUTCOMES:
Evaluate response rate, duration of response and progression free survival per RECIST criteria and the plasma and whole blood levels of quarfloxin. | One year

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Birmingham Hematology and Oncology, Birmingham, Alabama
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Ocala, Florida
  - Southern New Mexico Cancer Center, Las Cruces, New Mexico
  - Texas Oncology, Amarillo, Texas
  - Texas Oncology, Dallas, Texas
  - El Paso Cancer Treatment Center, El Paso, Texas
  - Cancer Care Centers of South Texas, Kerrville, Texas
  - UT Health Science Center, San Antonio, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Northwest Cancer Specialists, Vancouver, Washington